CLINICAL TRIAL: NCT02930980
Title: Micra Accelerometer Sensor Study 2
Acronym: MASS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MDT16023
Record Dates: First submitted 2016-10-06; First posted 2016-10-12 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Software (Experimental): Investigational Software loaded on Micra device
  Interventions: Device: Investigational Software loaded on Micra device

INTERVENTIONS:
Device: Investigational Software loaded on Micra device — Subject will receive an investigational software loaded on subject's Micra device

SUMMARY:
The purpose of the MASS2 is to characterize accelerometer signals of Micra implantable device during different postures and activities and to understand the source of the sensed motion, in order to test feasibility for future enhancements in device functionalities.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years old
* Subject is implanted with a Micra device
* Subject or witness (if applicable as per local regulation) is able and willing to provide Informed Consent

Exclusion Criteria:

* Subject is in atrial fibrillation
* Subject is not able to perform study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Kepler Universitätsklinikum, Linz, Austria
- France (2):
  - Hôpital cardiologique du Haut-Lévêque, Pessac
  - CHRU Tours - Hopital Trousseau, Tours
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chinitz L, Ritter P, Khelae SK, Iacopino S, Garweg C, Grazia-Bongiorni M, Neuzil P, Johansen JB, Mont L, Gonzalez E, Sagi V, Duray GZ, Clementy N, Sheldon T, Splett V, Stromberg K, Wood N, Steinwender C. Accelerometer-based atrioventricular synchronous pacing with a ventricular leadless pacemaker: Results from the Micra atrioventricular feasibility studies. Heart Rhythm. 2018 Sep;15(9):1363-1371. doi: 10.1016/j.hrthm.2018.05.004. Epub 2018 May 11. PMID 29758405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Software
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Software
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 14
  France | 20
  Spain | 9
Weight [Mean (Standard Deviation); unit: kg] | 76.5 (14.9)
Height [Mean (Standard Deviation); unit: cm] — Population: The difference between row population and overall is due to missing data.
  cm
    number analyzed (Participants) | 42
    (all) | 167 (10.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: The difference between row population and overall is due to missing data.
  kg/m^2
    number analyzed (Participants) | 42
    (all) | 27.6 (4.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Population: The difference between row population and overall is due to missing data.
  mm Hg
    number analyzed (Participants) | 42
    (all) | 138.9 (26.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Population: The difference between row population and overall is due to missing data.
  mm Hg
    number analyzed (Participants) | 41
    (all) | 76.2 (13.7)
Implant Duration [Mean (Standard Deviation); unit: days] | 369 (354)
Implant Location [Count of Participants; unit: Participants]
  RV Septum | 14
  RV Apex | 22
  RV Mid Septum | 7
Rhythm at time of software download [Count of Participants; unit: Participants]
  Sinus without 2nd or 3rd Atrioventricular block | 31
  Atrial Tachycardia (AT) | 1
  Atrial Fibrillation (AF) | 1
  Sinus with 2nd or 3rd Atrioventricular block | 10

OUTCOME MEASURES:

1. Primary Outcome: Waveform and Components of Accelerometer Signal
Description: Accelerometer signal was measured using the 3 axis Micra accelerometer (Vector 1 was labelled as V1, Vector 2 as V2, Vector 3 as V3).
  Components of the accelerometer signals (unit (g) represent acceleration)were identified and labelled as A1 (acceleration associated with ventricular systole), A2 (ventricular diastole), A3 (early passive filling), and A4 (active filling). The A4 signal is associated with atrial contraction and active filling.
Time Frame: For approximately two hours after software download
Population: Of the 43 subjects enrolled, 12 with Atrial tachycardia / Atrial fibrillation and 2nd degree or greater atrioventricular block were excluded from analysis since the A4 signal is absent or variable. An additional 4 subjects in sinus rhythm were excluded from analysis due to frequent pacing or telemetry noise, resulting in 27 subjects for analysis.
Measure: Mean (Standard Deviation); unit: g (unit (g) represent acceleration)
Arm/Group | Investigational Software
Number analyzed (Participants) | 27
g (unit (g) represent acceleration)
  A4 (g) in V1 | 0.15601 (0.08900)
  A4 (g) in V2 | 0.19222 (0.11058)
  A4 (g) in V3 | 0.14398 (0.08532)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected for each subject since subject enrollment until subject study exit (approx 2 hours).
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information, does not differ from the clinical trials.gov
Arm/Group | Investigational Software
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT02930980/Prot_SAP_000.pdf